CLINICAL TRIAL: NCT04476186
Title: The Effectiveness of Oral Acyclovir in the Treatment of Molluscum Contagiosum in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dalia Mahran (Other)
Collaborators: assistant professor Ghada M. Khafagy (Unknown); Dr. Marwa Diaaeldeen Abbass Hasan (Unknown); Prof. Dr. Emad Taha Abd-Elahim Ebiad (Unknown)
Responsible Party: Sponsor-Investigator, Dalia Mahran, professor of public health and community medicine, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: site of study assiut U H
Record Dates: First submitted 2020-07-06; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Active Comparator): 200 mg of oral acyclovir 5 timed per day for 5 days per week for maximum 1 month
  Interventions: Drug: Acyclovir
- controlled group (Placebo Comparator): KOH 10 % solution local application with apiece of cotton 2 time per day maximum for 1 month
  Interventions: Drug: KOH 10 %

INTERVENTIONS:
Drug: Acyclovir — oral syrp
  Other Names: Zovirax - Acyclovir
  Arms: treatment group
Drug: KOH 10 % — solution for local application
  Other Names: KOH
  Arms: controlled group

SUMMARY:
The investigators will study the effectiveness of acyclovir in the treatment of molluscum contagiosum in assiut university hospital - dermatological out patient clinic the treatment group will receive acyclovir 200 mg 5 times per day the controlled group will receive local KOH solution

DETAILED DESCRIPTION:
Study population:

Site of the study: The outpatient dermatological clinic in Assiut university hospital.

Participants: children (2 -16) years' old attending dermatological clinic in Assiut university hospital and their parents.

Methodology in details:

1. We will use the social media as " Facebook" to invite patient to visit the clinic and follow up them due to the protective measures of covid 19.
2. Diagnosis of the patient with molluscum contagiosum according to the clinical picture
3. Collecting data including personal and clinical data through interviewing the patient and his or her parents
4. Pictures of the lesions will be taken before and after treatment after patient consent.
5. We will Randomly assigning the patient to either treatment group or controlled group according to simple random table
6. Prescribing the treatment according to the patient group
7. Follow up of the patient after 1 weak and each week according to the response to treatment or presence of complication

Inclusion criteria:

Children (5 -15) years old with Molluscum contagiosum.

Exclusion criteria:

1. Molluscum contagiosum with Inflamed spot
2. Known immune compromised children
3. Molluscum lesion in the eye lid.
4. Children with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Children (2 -16) years old with Molluscum contagiosum.

Exclusion Criteria:

* Molluscum contagiosum with Inflamed spot Known immune compromised children Molluscum lesion in the eye lid. Children with renal impairment.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-29 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patient with complete clearance of all molluscum lesions. | 3 month for each participant
  we will measure the percentage of patient recovered from all lesion

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Mahmoud, Assist Prof, Principal Investigator — Cairo University
Locations (1):
- Hamdy Gomaa, Asyut, New Assiut City, Egypt

IPD SHARING:
Plan to Share IPD: No